CLINICAL TRIAL: NCT05508763
Title: Personalised Therapeutics @ Leiden University Medical Center
Brief Title: Personalised Therapeutics @LUMC
Acronym: PT@LUMC
Status: Active, not recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: bio.logis digital health GmbH (Unknown)
Responsible Party: Principal Investigator, J.J.Swen, Professor of Clinical Pharmacy and Pharmacogenetics, Leiden University Medical Center
Other Study IDs: NL78161.058.21
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Adverse Drug Reaction
Keywords: Pharmacogenetics
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PGx-guided dosing: This group will be genotyped for 14 pharmacogenes at the start of the study.
  Interventions: Genetic: Genetic test for 14 pharmacogenes
- Standard of care: This group will be genotyped for 14 pharmacogenes at the end of the study.

INTERVENTIONS:
Genetic: Genetic test for 14 pharmacogenes — Genotyping with the Global Diversity Array-8 v1.0 BeadChip with enhanced PGx
  Groups: PGx-guided dosing

SUMMARY:
In PT@LUMC 2000 patients will be randomized between a PGx-guided dosing group and a standard of care group. The patients will be followed for one year in which they will be asked to report adverse drug reactions at one, three, six and twelve months.

DETAILED DESCRIPTION:
Rationale: Pharmacogenomics (PGx) is the study of genetic variability affecting an individual's response to a drug. PGx is a critical component of personalized medicine. Currently, PGx is applied for individual drugs and/or individual genetic variants. Recently a pre-emptive panel-based approach was proposed including 48 PGx variants covering 13 genes for which the Dutch Pharmacogenetic Working Group (DPWG) has issued evidence based drug dosing guidelines. The PGx panel contains all genetic variants that are considered actionable by the DPWG i.e. requiring a dose adjustment or switch to another drug. Interestingly, more than 95% of the Dutch population carries one or more actionable genotype(s) for one of the genes covered by this panel and 10% carries 4 or more. Based upon national prescription data we estimate that 5.6% of all first prescriptions would require an individualization of the dose or drug. However, in current clinical practice the potential of PGx testing is not fully exploited and the impact for LUMC is unknown. Therefore a prospective study on pre-emptive PGx testing will be performed in the LUMC. In this study 2.000 patients will be randomized to PGx-guided dosing or standard of care.

In addition, we plan to conduct sub-studies with the obtained data. The first study aims to explore novel associations of genetic variants with variability in drug response. The second aims to explore the impact of concomitant medication and other non-genetic factors on pharmacogenetic associations in a pragmatic setting.

Primary objective: To implement pre-emptive panel based PGx testing in the LUMC and determine patient benefit of PGx guided drug prescription and dispensing.

Study design: A prospective, open, randomized study in 2,000 patients with a duration of 2 years.

Study population: Patients over 18 years old undergoing medication verification in the LUMC.

Study procedure: Patients are randomized to PGx-guided dosing or standard of care. The PGx-guided group receives pre-emptive PGx testing for a panel of 14 genes (including 227 PGx variants) followed by personalized drug and dose recommendations for newly prescribed drugs. Recommendations are based on the guidelines of the Dutch Pharmacogenetics Working Group. Patients in the control group will receive usual drug prescriptions, without PGx-guided drug or dose selection.

Main study parameters/endpoints: The primary outcome is the occurrence of drug-genotype associated adverse drug reactions (ADR) in the first 12 months following the genetic test. The outcome is dichotomized at ≥ grade 3 CTC-AE.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness. Participation in this study carries a small extra burden:

1) 10 ml additional blood will be collected during a venipuncture that is planned as part of regular treatment. 2) to complete an online questionnaires at one, three, six and twelve months. No extra visits to the clinic are necessary. Benefits to patients in the study arm include a potentially reduced risk of ADRs. All patients will receive their pharmacogenetic profile which can be used to individualize drug treatment based on the DPWG guidelines. Overall, minimal risks are expected for included patients due to the fact that all of the drugs included within this study have previously been licensed for routine use and thus have been evaluated as having a positive benefit/risk ratio. The DPWG guidelines are based on systematic review of the literature, have been published in peer-reviewed journals and are commonly accepted.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent (IC) prior to any study specific procedures.
* Be aged ≥18
* A venapunction as part of routine treatment
* Receive a medication verification interview
* Be able and willing to be followed-up for at least one year

Exclusion Criteria:

* Pregnancy or lactating
* Previous participation in the PREPARE trial (NCT03093818, NL60069.058.16)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of 18 years of age or older that participate in medication verification in the LUMC are eligible to participate.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
ADRs grade >3 total | One year
  The primary outcome will be the occurrence of clinically relevant (classified as NCI-CTCAE grade 3, 4, or 5) patient reported ADRs within one year of follow-up.

SECONDARY OUTCOMES:
ADRs grade >3 | One, three, six and twelve months
  The occurrence of clinically relevant (classified as NCI-CTCAE grade 3, 4, or 5) patient reported ADRs, attributable to a PGx drug, at one, three, six and twelve months of follow-up.
Acceptance to recommendations | One year
  Acceptance of the recommendations measured by comparing the number of dose adjustments and medication switches in the study and control arm.
Cost-effectiveness | One year
  The cost-effectiveness of a pre-emptive PGx panel test will be analysed by relating healthcare costs (including genetic testing, drugs and ADR-related care) to quality-adjusted life years (estimated using the EQ-5D-5L).
ADRs grade >2 total | One year
  The occurrence of clinically relevant (classified as NCI-CTCAE grade 2, 3, 4, or 5) patient reported ADRs, attributable to a PGx drug, within one year of follow-up.
ADRs grade >2 | One, three, six and twelve months
  The occurrence of clinically relevant (classified as NCI-CTCAE grade 2, 3, 4, or 5) patient reported ADRs, attributable to a PGx drug, at one, three, six and twelve months of follow-up.
Frequency of PGx drug prescriptions | One year
  The frequency of PGx drug prescriptions (per PGx gene) (corrected for dose changes due to PGx outcome) within one year of follow-up.

OTHER OUTCOMES:
The number of drugs per patient. | One year
The number of ADRs per patient ≥ grade 3. | One year
The number of ADRs per patient ≥ grade 2. | One year
The number of dose adjustment based on PGx guidelines. | One year
The total number of actionable PGx genes per patients. | One year
The total number of PGx drugs per patient. | One year
The treatment effectivity via routine drug levels (only those that are collected routinely) as a proxy for exposure. | One year
  Depending on the drug a different level (higher or lower) provides information regarding the treatment
Patient-reported drug adherence. | One year
  Drug adherence will be questioned during the study, the different moments will be compared and the overall drug adherence in the study will be addressed. A lower answer indicates less drug adherence and a higher score better drug adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No